CLINICAL TRIAL: NCT04668287
Title: Improving Students' Self-esteem With an Online Intervention Based on the Fennel Model: An Open-label, Uncontrolled Pilot Trial
Brief Title: Improving Students' Self-esteem With an Online Intervention
Acronym: SSEONI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West University of Timisoara (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WUTimisoara
Record Dates: First submitted 2020-12-08; First posted 2020-12-16 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-02

CONDITIONS: Self Esteem

STUDY DESIGN:
Intervention Model Description: Open-Label Pilot Study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Increasing Self-Esteem (Other): All participants will be included in working groups.
  Interventions: Behavioral: Increasing self-esteem

INTERVENTIONS:
Behavioral: Increasing self-esteem — During 5 weeks, participants will be part of one of the working groups in which they'll be taught by a counselor about how a low self-esteem develops and what have to be done for improving self-esteem, based on the Melanie Fennel' model.

SUMMARY:
The aim of this study is to measure the impact of an online intervention on students' self-esteem, using the model outlined by Melanie Fennell.

DETAILED DESCRIPTION:
The purpose of this study is to test the level of students' self-esteem (explicit and implicit) before and after an online intervention. All selected participants will enjoy one of the online working groups led by a psychologist for five weeks. In these group sessions, students will be trained to identify how their low self-esteem was developed, what are those factors that maintain their low self-esteem and what can they do for improving their low self-esteem, using Fennell model.

ELIGIBILITY:
Inclusion Criteria:

* Low Self-Esteem (Cut-off=35 at Rosenberg self-esteem scale)
* Being first year student in West University of Timisoara

Exclusion Criteria:

* Severe clinical depression symptoms (Cut-off=15 at PHQ9)
* Severe clinical anxiety symptoms (Cut-off=15 at GAD7)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Changes in Rosenberg's Self Esteem Scale | Change from Pre- to Post-Intervention (5 weeks)
  Rosenberg's Self Esteem Scale is a self-esteem measure widely used in social-science research. It is a ten-item likert-type scale with items answered on a four-point scale-from strongly disagree to strongly agree. The scale measures global self-worth by measuring both positive and negative feelings about the self. The minimum score of Rosenberg's Self Esteem Scale is 10 and the highest one is 40. A higher score means a better outcome.

SECONDARY OUTCOMES:
Name Letter Test | Change from Pre- to Post-Intervention (5 weeks)
  Name Letter Test is used to measure implicit self-esteem by testing the tendency to evaluate alphabetical letters in one's name, especially initials, particularly favorably.
Academic Burnout Scale | Change from Pre- to Post-Intervention (5 weeks)
  This scale is designed to measure the level of students' burnout. It contains 3 subscales: Exhaustion (minimum score: 5, maximum: 25), Cynicism (minimum score: 5, maximum: 25), Inefficacy (minimum score: 6, maximum: 30). A higher score means a worse outcome. Beside that, it can be scored Core Burnout, as sum between Exhaustion and Cynicism.
Generalised Anxiety Disorder Assessment (GAD7) | Change from Pre- to Post-Intervention (5 weeks)
  Generalised Anxiety Disorder Assessment is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. The minimum score of Generalised Anxiety Disorder Assessment is 0 and the highest one is 21. A higher score means a worse outcome (a higher level of anxiety).
Patient Health Questionnaire-9 (PHQ9) | Change from Pre- to Post-Intervention (5 weeks)
  Patient Health Questionnaire-9 was designed to measure participant's severity of depression using DSM IV criteria. The minimum score of Patient Health Questionnaire-9 is 0 and the highest one is 27. A higher score means a worse outcome (more severe symptoms of depression).
Treatment Satisfaction Questionnaire | Post-Intervention (5 weeks)
  Treatment Satisfaction Questionnaire is a scale designed to measure the level of students' satisfaction with intervention. The items refer to the content of the intervention, being open and close questions.
Therapeutic factors | Post-Intervention (5 weeks)
  A 9 item questionnaire designed to measure the impact of some of the therapeutic factors as universality, altruism, instillation of hope, etc (Yalom, I. D., & Leszcz, M. (Collaborator). (2005). The theory and practice of group psychotherapy (5th ed.)). For each of the 9 factors, the minimum score is 1 and the maximum one is 5. A higher score means a better outcome (that factor is relevant for intervention).
System usability | Post-Intervention (5 weeks)
  A 10 item questionnaire designed to measure participants' satisfaction with Zoom, the online platform used for weekly meetings. The minimum score of System Usability Scale is 10 and the highest one is 50. A higher score means a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- West University of Timișoara, Timișoara, Romania